CLINICAL TRIAL: NCT05912465
Title: The Role of 18F-FDG PET/CT in the Early Prediction of Cachexia in Lung Cancer Patients
Brief Title: Predicting Lung Cancer-Associated Cachexia With PET Imaging
Acronym: LUCAPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Leipzig (Other); Careggi Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Marcus Hacker, Head of the Division of Nuclear Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2091/2022
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cachexia; Lung Neoplasm
Keywords: Cancer cachexia; Positron emission tomography; Metabolic changes; Lung cancer; Muscle wasting; Computed tomography; Fluorodeoxyglucose F18; Organ connection
MeSH Terms: conditions — Cachexia; Lung Neoplasms; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: The overall model of this study involves enrolling a total of 150 patients from three different sites. These patients will undergo baseline PET/CT imaging to assess their metabolic changes, as well as provide clinical information through medical history review and physical examinations. Additionally, blood samples will be collected for laboratory tests, and patients will complete questionnaires to evaluate psychological stress levels. This comprehensive approach aims to gather a range of data including imaging, clinical information, blood biomarkers, and psychological assessments to investigate the relationship between cancer cachexia, stress, and metabolic changes in lung cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment-Naive Lung Cancer Patients (Experimental): This arm includes 150 treatment-naive lung cancer patients. Assessments include medical history, physical exams, lab tests, and imaging. Objective: investigate cancer cachexia, stress, and metabolic changes. Cachexia criteria: weight loss, reduced food intake, inflammation markers. Stress assessment: questionnaires, biomarkers. Metabolic changes measured by PET-CT scans analyzing FDG uptake in organs/lesions. Data will uncover the relationship between cancer cachexia, stress, and metabolic changes in treatment-naive lung cancer patients, leading to improved interventions/outcomes.
  Interventions: Other: Stress Reduction Training

INTERVENTIONS:
Other: Stress Reduction Training — A subgroup of patients from Vienna will undergo an additional PET/CT scan after the first follow-up PET/CT, which takes place one month after stress reduction training. The stress reduction training involves performing a breathing technique.

SUMMARY:
This prospective observational study aims to investigate the relationship between cancer cachexia, stress levels, and metabolic changes in 150 lung cancer patients. Cancer cachexia, characterized by weight loss and muscle wasting, significantly impacts patient outcomes. Psychological stress is thought to contribute to cachexia development. Assessments will include medical history, physical examinations, laboratory tests, and imaging. Cancer cachexia will be diagnosed based on weight loss, reduced food intake, and inflammation markers. Psychological stress will be evaluated using questionnaires and biomarkers. Metabolic changes will be assessed using positron emission tomography-computed tomography (PET-CT) scans. The primary objective is to determine differences in metabolic activity between cachectic and non-cachectic patients. Secondary objectives include evaluating changes in brain activity and exploring the relationship between stress, inflammation, and metabolism.

DETAILED DESCRIPTION:
Title: Investigation of the Relationship Between Cancer Cachexia, Stress, and Metabolic Changes in Lung Cancer Patients

Background: Cancer cachexia is a debilitating syndrome characterized by progressive weight loss, muscle wasting, and metabolic abnormalities. It significantly impacts patients' quality of life and survival outcomes. Psychological stress has been suggested as a potential contributor to cachexia development and progression. This study aims to investigate the association between cancer cachexia, stress levels, and metabolic changes in lung cancer patients.

Methods: This multicenter, prospective observational study will enroll 150 lung cancer patients. Eligible participants will undergo comprehensive assessments, including medical history review, physical examinations, laboratory tests, and diagnostic imaging. Cancer cachexia will be diagnosed based on established criteria, including weight loss, reduced food intake, and systemic inflammation markers. Psychological stress will be evaluated using validated questionnaires and stress biomarkers. Metabolic changes will be assessed through positron emission tomography-computed tomography (PET-CT) scans to measure fluorodeoxyglucose (FDG) uptake in organs and lesions.

Primary Objectives: The primary objective is to determine differences in FDG uptake between cachectic and non-cachectic lung cancer patients in various organs and lesions. Secondary objectives include evaluating changes in amygdalar FDG uptake after stress intervention and exploring the relationship between stress, inflammatory markers, and metabolic changes.

Statistical Analysis: Student's t-test will be used to compare FDG uptake between groups, and descriptive statistics will be calculated for each brain region. Sample size calculations indicate a need for approximately 30 subjects per group to detect significant differences. Data will be analyzed using appropriate statistical software.

Ethical Considerations: Informed consent will be obtained from all participants, and the study will adhere to the principles outlined in the Declaration of Helsinki and Good Clinical Practice guidelines. The study protocol has been submitted to the Ethics Committee and regulatory authorities for approval.

Conclusion: This study aims to provide insights into the relationship between cancer cachexia, stress, and metabolic changes in lung cancer patients. By investigating FDG uptake in different organs and lesions, as well as amygdalar FDG uptake before and after stress intervention, this research may contribute to the development of targeted interventions for cachexia management and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Confirmed diagnosis of lung cancer.
* Willingness to participate in the study and provide informed consent.
* Ability to comply with study procedures and follow-up visits.

Exclusion Criteria:

* Previous history of any other malignancy within the last 5 years, excluding non-melanoma skin cancer.
* Concurrent participation in another clinical trial involving an investigational product.
* Known contraindications or intolerance to PET/CT imaging or fluorodeoxyglucose (FDG).
* Presence of severe comorbidities that may interfere with study participation or affect the interpretation of results.
* Pregnant or lactating women, or those planning to become pregnant during the study period.
* Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Differences in FDG uptake (measured as SUVmean, max, min, peak) in organs, muscle, fat tissue between Cachectic and Non-Cachectic Lung Cancer Patients | F/U for 12 month minimum
  Measurement of fluorodeoxyglucose (FDG) uptake in various organs and lesions to characterize the metabolic differences between cachectic and non-cachectic lung cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hacker, Prof., Principal Investigator — Medical University of Vienna, Department of Radiology and Nuclear Medicine; Thomas Beyer, Prof., Principal Investigator — Medical University of Vienna, Center for Medical Physics and Biomedical Engineering; Osama Sabri, Prof., Principal Investigator — University of Leipzig Medical Center; Roberto Sciagrà, Prof., Principal Investigator — Careggi University Hospital
Locations (3):
- Medical University of Vienna, Vienna, Austria
- University of Leipzig Medical Center, Leipzig, Germany
- AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shiyam Sundar LK, Yu J, Muzik O, Kulterer OC, Fueger B, Kifjak D, Nakuz T, Shin HM, Sima AK, Kitzmantl D, Badawi RD, Nardo L, Cherry SR, Spencer BA, Hacker M, Beyer T. Fully Automated, Semantic Segmentation of Whole-Body 18F-FDG PET/CT Images Based on Data-Centric Artificial Intelligence. J Nucl Med. 2022 Dec;63(12):1941-1948. doi: 10.2967/jnumed.122.264063. Epub 2022 Jun 30. PMID 35772962
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- See also: Project Website — https://www.meduniwien.ac.at/web/en/forschung/projekte/lucapet/lucapet/